CLINICAL TRIAL: NCT06628141
Title: Enhancing Quality of Life in Cancer Patients Through Tailored Nutrition Support: a Comprehensive Approach
Acronym: BLOOMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UOMi Cancer Center (Other)
Collaborators: Dexeus Clinic Woman (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UOMi Cancer Center
Record Dates: First submitted 2023-11-22; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nutritional support tool (Experimental)
  Interventions: Other: Nutritional support tool

INTERVENTIONS:
Other: Nutritional support tool — Nutritional support tool

SUMMARY:
The study aims to investigate the impact of a dedicated nutritional assistance tool on patients with cancer and to measure its effects on several proposed indicators.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by cancer, who decided to participate to the study, signed the informed consent and whose life expectancy is higher than 1 (one) year.

Exclusion Criteria:

* Patients with an eating disorder of psychiatric or psychological origin, diagnosed before cancer treatment.
* Any other exclusion criteria as determined by the oncologist based on the patient's ability to successfully complete the program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Outcome Measure: Dietary Adherence | 1 year
  Dietary adherence will be measured by comparing the planned recipes provided to participants with the meals they report consuming each week. Participants receive 21 recipe suggestions (7 breakfasts, 7 lunches, 7 dinners) via a mobile app. The following tools and methods will assess adherence:
  Mobile Application Tracking: The app tracks participants' views of recipes and ingredient purchases via the integrated shopping list.
  Weekly Questionnaire: A self-reported questionnaire asks if participants:
  Followed the recipes using ingredients purchased via the app. Prepared recipes with their own ingredients. Ate meals not included in the plan. Adherence Calculation: Adherence is calculated as the ratio of recipes followed (via app or self-preparation) to the total number of recommended recipes (21 per week), expressed as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- UOMI Cancer Center Clínica Mi Tres Torres, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided